CLINICAL TRIAL: NCT03610217
Title: Pragmatic Clinical Trials in Scleroderma
Acronym: PCTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of West London (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Andreu Fernandez Codina, Principal investigator, University of Western Ontario, Canada
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 111419
Record Dates: First submitted 2018-07-25; First posted 2018-08-01 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Scleroderma, Systemic; Sclerosis, Systemic
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- Interstitial lung disease induction (Experimental)
  Interventions: Other: Interstitial lung disease induction algorithm
- Pulmonary arterial hypertension (Experimental)
  Interventions: Other: Pulmonary arterial hypertension algorithm
- Raynaud's phenomenon (Experimental)
  Interventions: Other: Raynaud's phenomenon algorithm
- Digital ulcers (Experimental)
  Interventions: Other: Digital ulcer algorithm
- Inflammatory arthritis (Experimental)
  Interventions: Other: Inflammatory arthritis algorithm
- Gastroesophageal reflux (Experimental)
  Interventions: Other: Gastroesophageal reflux algorithm
- Bacterial overgrowth (Experimental)
  Interventions: Other: Bacterial overgrowth algorithm
- Constipation (Experimental)
  Interventions: Other: Constipation algorithm
- Skin involvement (Experimental)
  Interventions: Other: Skin involvement algorithm
- Pain (Experimental)
  Interventions: Other: Pain algorithm

INTERVENTIONS:
Other: Interstitial lung disease induction algorithm — Patients failing first line mycophenolic acid (MFA) will be randomized to MFA plus rituximab or intravenous cyclophosphamide. If they fail the second line they will be crossed over to the other option.
  Arms: Interstitial lung disease induction
Other: Pulmonary arterial hypertension algorithm — Patients diagnosed with pulmonary arterial hypertension secondary to systemic sclerosis will be randomized to receive anticoagulation (warfarin, rivaroxaban or apixaban)
  Arms: Pulmonary arterial hypertension
Other: Raynaud's phenomenon algorithm — Patients with mild Raynaud's phenomenon not responding to the first line treatment (nifedipine), will be randomized to receive losartan or nifedipine plus atorvastatin or nifedipine plus losartan. If they fail the second line they will be crossed over to the other options randomly.
  Patients with severe Raynaud's phenomenon not responding to the first line treatment (nifedipine) or failing the previous mild Raynaud's algorithm, will be randomized to receive nifedipine plus sildenafil or nifedipine plus intravenous iloprost. If they fail the second line they will be crossed over to the other option.
  Arms: Raynaud's phenomenon
Other: Digital ulcer algorithm — Patients with active digital ulcers not healing after 3 months or developing new ones with nifedipine will be randomized to nifedipine plus sildenafil or nifedipine plus intravenous iloprost. If they fail the second line they will be crossed over to the other option.
  Patients who develop new digital ulcers under treatment with nifedipine will be randomized to nifedipine plus atorvastatin plus standard of care or nifedipine plus standard of care. If they fail the second line they will be crossed over to the other option.
  Arms: Digital ulcers
Other: Inflammatory arthritis algorithm — Patients with inflammatory arthritis failing methotrexate and/or prednisone and/or hydroxychloroquine and/or sulfasalazine will be randomized to receive intravenous rituximab or subcutaneous tocilizumab. If they fail the second line they will be crossed over to the other option.
  Arms: Inflammatory arthritis
Other: Gastroesophageal reflux algorithm — Patients with gastroesophageal reflux failing standard doses of proton pump inhibitors (PPI) will be randomized to receive double doses of PPI or standard dose of PPI plus ranitidine or double doses of PPI plus domperidone or double doses of PPI plus prucalopride/erythromycin. If they fail the second line they will be crossed over to the other options randomly.
  Arms: Gastroesophageal reflux
Other: Bacterial overgrowth algorithm — Patients with bacterial overgrowth will be randomized to receive erythromycin or metronidazole or amoxicillin. If they fail the second line they will be crossed over to the other options randomly.
  Arms: Bacterial overgrowth
Other: Constipation algorithm — Patients with constipation will be randomized to receive bisacodyl or magnesium sulphate or polyethylene glycol or senna.If they fail the second line they will be crossed over to the other options randomly.
  Arms: Constipation
Other: Skin involvement algorithm — Patients with skin involvement and modified Rodnan skin score <32 will be randomized to receive methotrexate or mycophenolic acid or methotrexate plus mycophenolic acid. If they fail the second line they will be crossed over to the other option.
  Patients with skin involvement and modified Rodnan skin score >32 will be randomized to receive methotrexate plus mycophenolic acid or intravenous cyclophosphamide. If they fail the second line they will be crossed over to the other option.
  Arms: Skin involvement
Other: Pain algorithm — Patients with pain failing first line treatment with acetaminophen or celecoxib or ibuprofen will be randomized to receive pregabalin or duloxetine. Patients with skin involvement and modified Rodnan skin score <32 will be randomized to receive methotrexate or mycophenolic acid or methotrexate plus mycophenolic acid. If they fail the second line they will be crossed over to the other option. In case they fail the second line they will be treated with medical marijuana.
  Arms: Pain

SUMMARY:
Systemic Sclerosis (SSc) is an autoimmune connective tissue disease characterized by autoantibodies, fibrosis and microvascular injury and endothelial cell activation that results in vascular damage. Vascular injury induces both innate and acquired immune responses resulting in fibroblast activation and organ fibrosis. SSc may target multiple organs, including: skin, lungs, heart, vascularization, kidneys, the gastrointestinal tract and musculoskeletal structures. Mortality among scleroderma patients is significant, with a 3.5 standardized mortality ratio (SMR) in studies of prevalent cases. This mortality may be increased in the early years of the disease, reaching a SMR of 4 in a multinational inception cohort. In general, treatment strategies target involved organs as early as possible to avoid damage. Many treatment options are available for each manifestation, but evidence with respect to the order of treatment is scarce. Financial costs, the lack of proper outcome measures, difficulty to recruit patients as a rare disease, all prevent the development of new big clinical trials, oppositely to other common diseases such as stroke or cancer. The heterogeneous features of SSc may make trials challenging. The current guidelines available are the British guidelines (2017) , and the updated European League Against Rheumatism (EULAR) guidelines, published in 2017. Management guidelines have some gaps regarding second-line treatment, combinations and there are no proposed algorithms.

With the pragmatic trials, the investigators intend to fill the gap between the complicated randomized clinical trials and the observational studies. Using the treatments that have already been proved useful in SSc, in an open-label randomized way and based on some refined expert-made algorithms, will allow the investigators to establish the order in how to use them.

Patients will be offered to participate with the collection of their clinical data and, if they give their consent, they will be randomized according to the algorithms. There will be an optional part of the study consisting in the collection of blood samples and skin samples for future research.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with an age >18 years meeting the 2013 SSc classification criteria managed at the Rheumatology division, St. Joseph's Healthcare London.
* Patients who refuse to be randomized for treatments but wish to provide their data for the registry will also be included, after signing the informed consent form.

Exclusion Criteria:

* Refusal to participate or to sign an informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Forced vital capacity % | 1 year
  Variation of the forced vital capacity %
Bleeding | 1 year
  Documentation of bleeding
Raynaud's phenomenon visual analog scale | 3 months
  Raynaud's phenomenon visual analog scale variation ranging from 0 to 100 mm (0 no Raynaud's phenomenon, 100 very intense Raynaud's phenomenon)
Time to the healing of a digital ulcer | 1 year
  Time to the healing of a digital ulcer
Time to the development of a new digital ulcer | 1 year
  Time to the development of a new digital ulcer
Disease activity score 28 | 3 months
  Disease activity score 28 accounting for tender and swollen joints over 28 possible joints. Values <2.6 remission, values <3.2 low disease activity, values >5.1 high disease activity
GERD-HRQL | 3 months
  Variation of the Gastro-esophageal reflux disease-health related quality of life questionnaire, ranging from 0 (no symptoms) to 75 (worst symptoms)
Diarrhea visual analog scale | 3 months
  Diarrhea visual analog scale variation ranging from 0 to 100 mm (0 no diarrhea, 100 very intense diarrhea)
Constipation visual analog scale | 3 months
  constipation visual analog scale variation ranging from 0 to 100 mm (0 no constipation, 100 very intense constipation)
Modified Rodnan skin score | 1 year
  Modified Rodnan skin score variation. Ranging from a total of 0 (no induration) to 51 (maximum induration)
Pain visual analog scale | 3 months
  Pain visual analog scale variation, ranging from 0 to 100 mm (0 no pain, 100 very intense pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Joseph's Health Care London, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fernandez-Codina A, Walker KM, Pope JE; Scleroderma Algorithm Group. Treatment Algorithms for Systemic Sclerosis According to Experts. Arthritis Rheumatol. 2018 Nov;70(11):1820-1828. doi: 10.1002/art.40560. Epub 2018 Sep 17. PMID 29781586
- See also: Related Info — https://www.sjhc.london.on.ca/rheumatology